CLINICAL TRIAL: NCT04084600
Title: The Effects of Manual Therapy on Chronic Pain and Functionality of Breast Cancer Survivors: a Randomized Controlled Trial
Brief Title: Effects of Manual Therapy on Chronic Pain and Functionality of Breast Cancer Survivors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study had to be stopped due to the COVID-19 pandemic. The University has been closed since the beginning of the pandemic until the present date (02/2021) due to the social distance imposed by the government.
Sponsor: University of the State of Santa Catarina (Other)
Responsible Party: Principal Investigator, Gilmar Moraes Santos, PT, Clinical Professor, University of the State of Santa Catarina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Manual Therapy BCS
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Medicine, Thai Traditional

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Once a week for 6 consecutive weeks, this group will receive a manual therapy protocol with an approach based on Taylor et al., 1990; Schleip et al., 2012; Bienfait, 1999 and Myers, 2016, lasting 20 minutes, focused on the upper quadrant homolateral to the surgery. Shortly thereafter, this group will participate in a kinesiotherapy protocol with stretching, mobility and strengthening exercises, also for 20 minutes. All sessions will be individual.
  Interventions: Other: Kinesiotherapy Protocol; Other: Manual Therapy Protocol
- Sham Group (Sham Comparator): Once a week for 6 consecutive weeks, this group will receive a soft and shallow traditional massage, lasting 20 minutes. Shortly thereafter, this group will participate to the same kinesiotherapy protocol with stretching, mobility and strengthening exercises, also for 20 minutes. All sessions will be individual.
  Interventions: Other: Kinesiotherapy Protocol; Other: Traditional Massage

INTERVENTIONS:
Other: Kinesiotherapy Protocol — Kinesiotherapy Protocol is an specific exercise based treatment designed to strengthening, gaining range of motion and stretching the muscles.
Other: Manual Therapy Protocol — Manual therapy protocol: is a manual treatment intended to the release of fascias and soft tissues.
  Arms: Intervention Group
Other: Traditional Massage — Traditional Massage is a gentle and superficial massage.
  Arms: Sham Group

SUMMARY:
the aim of this study is to verify whether manual therapy associated with kinesiotherapy is more effective than kinesiotherapy alone in the treatment of chronic pain and upper limb dysfunction in women surviving cancer of mama. It is a randomized controlled double blind clinical trial (evaluator and patient), parallel in two groups (Intervention Group and Sham Group). The intervention will last 6 weeks and chronic pain and upper limb functionality will be evaluated. Both groups will undergo a kinesiotherapy program once a week for 6 consecutive weeks. Also, participants in the intervention group will receive, once a week, a manual therapy protocol, while participants in the Sham group will receive traditional massage. Manual therapy associated with kinesiotherapy is expected to yield superior results to the isolated kinesiotherapy in chronic pain and upper limb functionality.

DETAILED DESCRIPTION:
This study will be a double-blind randomized controlled trial, parallel in two groups (intervention group and sham). Participants will initially be evaluated by a trained investigator who will be blinded and assigned randomly (random numbers generated on the computer) block for the intervention and sham groups by an opaque envelope draw. Participants will be randomized into two groups: intervention and sham. Both groups will undergo a kinesiotherapy program once a week for 6 consecutive weeks.

Also, participants in the intervention group will receive, once a week, a manual therapy protocol, while participants in the Sham group will receive traditional massage. When making the invitation to participate in the survey, individuals will not be required to participate if they do not agree, and therefore will not be penalized. Participants who agree to participate in the survey will sign a Free and Informed Consent Form and will be informed of the possibility of withdrawing from the survey at any stage, without penalty. The collection of the evaluation and intervention will be carried out in a salon Clinic School of Physiotherapy in the Center of Health and Sports Sciences (CEFID) of the State University of Santa Catarina (UDESC) in the city of Florianópolis- SC. All personal identification data of the participants will be preserved according to resolution of the national health council, taking into account the possibility of scientific dissemination of the results obtained. The risks of these procedures will be medium, since the participant may present muscle pain after the intervention protocol. To minimize these risks will be available, if necessary, attendance at the Clinic School of Physiotherapy. The sample will be selected in a non-probabilistic way for convenience. This study will include women diagnosed with breast cancer who have undergone breast surgery with curative intent and who have completed chemotherapy and / or radiotherapy treatments.

ELIGIBILITY:
Inclusion Criteria:

* age over 18 years;
* have had surgery to treat breast cancer;- have completed chemotherapy and / or radiotherapy;
* have upper quadrant pain homolateral to surgery for at least the last 3 months, with a score of 4 or more on the visual analog scale (VAS) in the last week
* present a score greater than or equal to 30 on the Arm, Shoulder, and Hand Dysfunction Questionnaire (DASH).

Exclusion Criteria:

* difficulty in understanding the Portuguese language to answer the questionnaires;
* have had bilateral surgery to treat breast cancer;
* be in palliative care;
* pregnant women;
* be using analgesic and / or anti-inflammatory drugs
* women with rheumatic diseases
* be in physical therapy during the intervention period.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

PRIMARY OUTCOMES:
Change in Chronic Pain Intensity | Change from Pre Intervention Chronic Pain Intensity at 6 weeks Post Intervention
  Chronic pain intensity will be evaluated through the analogue visual scale. It consists of a numbered line from 1 to 10, 0 being no pain and 10 the worst pain imaginable.
Change in Pain Location | Change from Pre Intervention Pain Location at 6 weeks Post Intervention
  Pain location will be assessed using a Body Pain Diagram. It is a graphical representation of a woman's body in anterior, posterior, and lateral views to identify the location and frequency of pain. In this diagram, women should mark with a X their main pain points in the upper quadrant homolateral to the surgery.
Change in Neuropathic Pain | Change from Pre Intervention neuropathic pain at 6 weeks Post Intervention
  Neuropathic Pain will be assessed using the Douler Neuropathique 4 Questionnaire. It aims to discriminate neuropathic pain from nociceptive pain. It consists of 10 items grouped into 4 sections. The first 7 items are related to pain quality (burning, painful cold, and electric shock) and its association with abnormal sensations (tingling, numbness, and itching). The remaining 3 items are associated with neurological examination in the painful area (touch hypoesthesia, needle stick hypoesthesia, and tactile allodynia). Each positive item receives a 1-point score and the total score is calculated as the sum of all 10 items. A score of 4 or higher indicates the diagnosis of neuropathic pain.
Change in central sensitization pain | Change from Pre Intervention central sensitization pain at 6 weeks Post Intervention
  Central sensitization pain will be assessed using the the Central Sensitization Questionnaire. It aims to evaluate the symptoms considered associated with central sensitization pain. The total score ranges from 0 to 100 and a score of 40 or more indicates the presence of central sensitization pain.
Change in pain dimensions | Change from Pre Intervention pain dimensions at 6 weeks Post Intervention
  Pain dimensions will be assessed using the McGill Pain Questionnaire. It is an instrument that assesses pain dimensions in physical (sensitive and discriminative) aspects, pain interpretation (affective and motivational) and pain understanding (cognitive and evaluative). It is made up of 4 large groups, divided into 20 smaller groups of words, each of which is related to a type of pain. The groups are numbered according to intensity, with 1 being the smallest: 10 groups of 42 words related to physical aspects; 5 groups of 14 words related to the affective part; 1 group of 5 words about pain in general; 4 groups of 17 words that did not fit the other groups, called miscellaneous. The values are summed and the result is given by the pain index (sum of the intensity values of the chosen descriptors, with a maximum value of 78) and by the number of descriptors (how many words were marked, with a maximum value of 20).

SECONDARY OUTCOMES:
Upper limb functionality | Change from Pre Intervention Upper limb functionality at 6 weeks Post Intervention
  The Arm, Shoulder and Hand Dysfunctions Questionnaire (DASH) will be used to assess disabilities and physical symptoms of the upper limbs. It is a 30-item questionnaire that evaluates the physical disabilities and symptoms of upper limbs in a wide variety of musculoskeletal disorders. The Likert score ranges from 1 to 5 and the total score ranges from 0 to 100, where higher scores represent higher physical disabilities and upper limb symptoms. The questions refer to the last week and the questionnaire items are divided into physical function, symptoms and social function.Questionnaire.
Muscle strength | Change from Pre Intervention Muscle strength at 6 weeks Post Intervention
  Muscle strength will be assessed by the Kendall scale, graded from 1 to 5.
Range of motion | Change from Pre Intervention Range of motion at 6 weeks Post Intervention
  The range of motion will be evaluated by a goniometer
Circumference of the arm | Change from Pre Intervention Circumference of the arm at 6 weeks Post Intervention
  The circumference of the arm will be evaluated by the perimeter.

CONTACTS AND LOCATIONS:
Overall Officials: Gilmar M Santos, PhD, Study Chair — Universidade do Estado de Santa Catarina this account disabled
Locations (1):
- Santa Catarina State University, Florianópolis, Santa Catarina, Brazil